CLINICAL TRIAL: NCT06560944
Title: Effects of Oral Contraceptive Consumption Timing on Cognition and Metabolism
Brief Title: Oral Contraceptive Consumption Timing and Cognition and Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lincoln (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 718
Record Dates: First submitted 2023-06-27; First posted 2024-08-19 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Cognitive Change
MeSH Terms: interventions — Contraceptives, Oral, Combined

STUDY DESIGN:
Intervention Model Description: Randomised-controlled crossover trial
Who Masked: Participant, Investigator
Masking Description: Random number generator, via technicians, concealed allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral contraceptive (Experimental): Participants existing oral contraceptive to be ingested at 8am on a day between 3 to 21 of pill consumption. Placebo consumed ~2 hours later
  Interventions: Drug: Combined oral contraceptive pill
- Placebo (Placebo Comparator): Placebo ingested at 8am on a day between 3 to 21 of pill consumption. Participants existing oral contraceptive consumed ~2 hours later
  Interventions: Drug: Combined oral contraceptive pill

INTERVENTIONS:
Drug: Combined oral contraceptive pill — Ingesting their existing combined oral contraceptive pill at a specific time of day in relation to assessment of outcome measures

SUMMARY:
The aim of this randomised-controlled trial is to examine whether the timing of oral contraceptive administration affects cognitive function, substrate metabolism and exercise performance.

Participants will attend the laboratory for a familiarisation session, followed by two main trials in which cognition and exercise metabolism and performance are measured. In one trial they will be given their oral contraceptive 60 minutes before testing begins, in the other they will be given a placebo. Following testing (~60 minutes), participants will consume the alternative pill.

DETAILED DESCRIPTION:
Reproductive hormones, such as oestrogen and progesterone, are known to affect cognitive function (i.e. thinking, learning and processing information) and substrate metabolism (i.e. how the body uses carbohydrates and fats). Oral contraceptives contain synthetic versions of reproductive hormones and are used by approximately half of women of reproductive age. When oral contraceptives are ingested, the concentrations of these synthetic hormones spike in the blood for several hours, yet no research has explored the effect of this spike on how the body works, especially with regards to cognitive function and substrate metabolism. If this spike in synthetic hormone concentrations affects cognition or metabolism, this could influence the way in which women use oral contraceptives, such as altering the timing of ingestion to improve performance and health outcomes.

The proposed study will use participants that currently use a specific preparation of oral contraceptive (30micrograms ethinyl estradiol and 150mg Levonorgestrel) and compare cognitive function and substrate metabolism on an occasion when a placebo is consumed (lactose - no hormones), to an occasion when their oral contraceptive is consumed. It takes approximately 60-90 minutes for concentrations of hormones to peak in the blood following ingestion, therefore measurements of cognitive function and substrate metabolism will be taken at this time. Cognitive function will be measured using a battery of tests administered orally or via a laptop and substrate metabolism will be measured by collecting expired air via a mouthpiece at rest and during exercise on a treadmill, during which time perceived difficulty of the exercise (rate of perceived exertion) and feelings (felt arousal) will be measured. Venous blood samples will be drawn at baseline (immediately before consumption of first pill/placebo) and 90 minutes following this. The participants will consume either the placebo or oral contraceptive (whichever was not initially consumed) following the testing protocol to ensure that their contraceptive protection is maintained.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 18-35 years
* The use of the same oral contraceptive (30 micrograms ethinyl estradiol and 150mg levonorgestrel) for at least 6 months
* Physically active and able to take part in treadmill-based exercise
* Speak fluent English

Exclusion Criteria:

* Use of any other type of hormonal contraception
* Aged < 18 or > 35 years
* Poly-cystic ovarian syndrome
* Endometriosis
* Pregnant
* Child birth or lactation in the previous 6 months
* Body mass index < 18.5 or > 30 kg.m2
* Any disorder known to affect metabolic health
* History of head injury/neurological disorders
* Use of any steroid-based medication or medications known to influence the central nervous system
* History of psychiatric disorders such as major depression or an anxiety disorder
* Smokers
* Suffer from (or have suffered from) a heart complaint
* Advised by medical professional to refrain from high intensity exercise
* Current muscle or joint injury

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
Rey Auditory Verbal Test Performance | 60-90 minutes post oral contraceptive/placebo ingestion
  Acquisition, Learning rate, Proactive Interference, Retroactive interference, Forgetting
Mental Rotation test | 60-90 minutes post oral contraceptive/placebo ingestion
  Accuracy, Response time
Verbal Fluency | 60-90 minutes post oral contraceptive/placebo ingestion
  Words said
Stroop test | 60-90 minutes post oral contraceptive/placebo ingestion
  Accuracy, Response time
Corsi blocks | 60-90 minutes post oral contraceptive/placebo ingestion
  Correct sequences, longest sequence
Rapid Visual Information Processing | 60-90 minutes post oral contraceptive/placebo ingestion
  Proportion correct, Response time
Rating of perceived exertion | During final minute of of 6 minutes exercise at both 70 and 90% lactate threshold. Exercise takes place approximately 90 minutes post oral contraceptive/placebo ingestion
  Borg rating of perceived exertion (RPE) scale from 6-20. Higher value indicates greater exertion
Felt arousal | During final minute of of 6 minutes exercise at both 70 and 90% lactate threshold. Exercise takes place approximately 90 minutes post oral contraceptive/placebo ingestion
  Felt arousal scale from 1-6. Higher value indicates greater level of arousal
Feeling scale | During final minute of of 6 minutes exercise at both 70 and 90% lactate threshold. Exercise takes place approximately 90 minutes post oral contraceptive/placebo ingestion
  Feeling scale -5 to +5. Higher value indicates more positive feeling.
Heart rate | During final minute of of 6 minutes exercise at both 70 and 90% lactate threshold. Exercise takes place approximately 90 minutes post oral contraceptive/placebo ingestion
  beats per minute
Carbohydrate oxidation | During final minute of of 6 minutes exercise at both 70 and 90% lactate threshold. Exercise takes place approximately 90 minutes post oral contraceptive/placebo ingestion
  Rate of carbohydrate use
Fat oxidation | During final minute of of 6 minutes exercise at both 70 and 90% lactate threshold. Exercise takes place approximately 90 minutes post oral contraceptive/placebo ingestion
  Rate of fat use
Respiratory exchange ratio | During final minute of of 6 minutes exercise at both 70 and 90% lactate threshold. Exercise takes place approximately 90 minutes post oral contraceptive/placebo ingestion
  Ratio of carbohydrate and fat metabolism
Breathing frequency | During final minute of of 6 minutes exercise at both 70 and 90% lactate threshold. Exercise takes place approximately 90 minutes post oral contraceptive/placebo ingestion
  breaths per minute
Maximal oxygen consumption (VO2max) | During maximal exercise test which occurs approximately 110 minutes post oral contraceptive/placebo ingestion
  Maximal rate of oxygen used
Time to exhaustion | During maximal exercise test which occurs approximately 110 minutes post oral contraceptive/placebo ingestion
  Time before test termination
Maximal heart rate | During maximal exercise test which occurs approximately 110 minutes post oral contraceptive/placebo ingestion
  Maximal heart rate achieved

SECONDARY OUTCOMES:
Seum ethinyl estradiol | Baseline and immediately post cognitive function tests
  Synthetic oestrogen concentrations in blood
Serum Levonorgestrel | Baseline and immediately post cognitive function tests
  Synthetic progesterone concentrations in blood

CONTACTS AND LOCATIONS:
Overall Officials: Dan Martin, PhD, Principal Investigator — University of Lincoln
Locations (1):
- Dan Martin, Lincoln, Lincolnshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No